CLINICAL TRIAL: NCT06206798
Title: The Effects of Resourcefulness Group Intervention on Recovery and Quality of Life in Patients With Chronic Schizophrenia.
Brief Title: Resourcefulness Group Intervention on Recovery and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Huaining Kao, graduate student, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C110142
Record Dates: First submitted 2023-08-09; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Chronic Schizophrenia; Quality of Life; Recovery
Keywords: Resourcefulness; Chronic Schizophrenia; Resourcefulness Group; Recovery; Quality of Life

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 1. Subjects were randomly assigned to the experimental or the control group.
  2. There were 20 members in the experimental group who received 6-week intervention activities.
  3. Each subject was asked to fill out the questionnaires three times in total. The first time was before the intervention; the second time was right after the intervention; and the last time was four weeks later of the intervention.
  Interventions: Behavioral: Resourcefulness Group
- control group (No Intervention): 1. There were 20 members in the control group who accepted chronic nursing care as usual without any nursing intervention.
  2. Each subject was asked to fill out the questionnaires three times in total. The first time was the same time as the experimental group; the second time was 6 weeks after the first test; and the last time was four weeks after the second test.

INTERVENTIONS:
Behavioral: Resourcefulness Group — The content of the Resourcefulness intervention group includes 6 sessions such as session 1 to introduce resourcefulness skills; sessions 2-4 to discuss personal resourcefulness skills including planning daily activities, and positive self-talk; sessions 4-5 to discuss social resourcefulness skills including relying on family or friends, and seeking professional assistance.
  Arms: experimental group

SUMMARY:
The purpose of this study was to test the effects of resourcefulness group intervention on facilitating recovery and improving the quality of life in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
Purpose: This study aimed to explore the effects of resourcefulness group intervention on facilitating recovery and improving the quality of life in patients with chronic schizophrenia.

Methods: A longitudinal and interventional study with a quasi-experimental research design and convenience sampling were used in this study. Patients with chronic schizophrenia from a psychiatric hospital in northern Taiwan were recruited as subjects and were divided under random assignment into the experimental group and the control group with twenty participants in each. The twenty participants in the experiment group were further randomly distributed into two groups. Both received resourcefulness group intervention weekly for six weeks, while the control group followed regular care routines and underwent conventional treatment. All participants took a pretest before the intervention, the first posttest after six rounds of intervention, and the second posttest four weeks after the group intervention was completed. Data were collected using structured questionnaires, including the Chinese version of the Resourcefulness Scale (C-RS), the Chinese Questionnaire about the Process of Recovery (QPR), the WHOQOL-BREF Taiwan Version, and other personal information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been diagnosed with schizophrenia by a psychiatrist for more than two years and are currently receiving rehabilitation treatment in a chronic ward.
* Age between 20-64 years old.
* Those with stable conditions can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* Exclude clients with Intellectual Disabilities, Organic Encephalopathy, Substance-related and addictive disorders, Personality disorders, Dementia, Cancers, etc.
* Those who are unable to understand the contents of the consent form.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Chinese version of Resourcefulness Scale | Up to 10 weeks. The pre-test questionnaire will be completed before the group starts, the first post-test will be administered after the group, and the second post-test will be administered 4 weeks after the group ends
  Resourcefulness
Chinese questionnaire about the process of recovery | Up to 10 weeks. The pre-test questionnaire will be completed before the group starts, the first post-test will be administered after the group, and the second post-test will be administered 4 weeks after the group ends
  recovery
WHOQOL-BREF Taiwan version | Up to 10 weeks. The pre-test questionnaire will be completed before the group starts, the first post-test will be administered after the group, and the second post-test will be administered 4 weeks after the group ends
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Chien Yu Lai, PhD., Study Director — Associate professor
Locations (1):
- Peihsin Hospital, New Taipei City, Tamsui Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No